CLINICAL TRIAL: NCT03374917
Title: An Open-Label Study in Subjects With Parkinson's Disease to Evaluate the Safety and Tolerability of Titration and Continuous Subcutaneous Infusion of ABBV-951 for up to 4 Weeks in an Outpatient Environment
Brief Title: A Study in Subjects With Parkinson's Disease to Evaluate the Safety and Tolerability of Titration and Continuous Subcutaneous Infusion of ABBV-951 in an Outpatient Environment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-739
Record Dates: First submitted 2017-12-08; First posted 2017-12-15 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Parkinson's Disease (PD)
Keywords: carbidopa; levodopa
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABBV-951 (Experimental): ABBV-951 administered by continuous subcutaneous infusion (CSCI) for 4 weeks.
  Interventions: Drug: ABBV-951

INTERVENTIONS:
Drug: ABBV-951 — powder for solution

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of 4 weeks of continuous infusion with ABBV-951 in adult subjects with Parkinson's Disease (PD).

ELIGIBILITY:
Inclusion Criteria:

* Subject with a diagnosis of definite idiopathic Parkinson's disease (PD) that is levodopa-responsive according to the United Kingdom Parkinson's Disease Society Brain Bank Criteria.
* Subject must be taking an optimized and stable regimen of oral medications for PD, which has remained stable and unchanged for at least 30 days before enrollment in this study.
* Subject is judged inadequately controlled on current therapy in the opinion of the Investigator and must experience a minimum of 2.5 hours of "off" time per day prior to Enrollment.
* Subjects with a MMSE score greater than or equal to 24 and considered by the Investigator to not have dementia.

Exclusion Criteria:

* Subjects with clinically significant electrocardiogram (ECG) values.
* History of significant skin conditions or disorders that in the Investigator's opinion would interfere with the infusion of the study drug or could interfere with study assessments.
* Receipt of an investigational product within at least 6 weeks prior to study drug administration.
* Subjects with moderate to severe kidney disease.
* Consideration by the investigator for any reason that the subject is an unsuitable candidate to receive ABBV-951.
* Patient/caregiver that cannot demonstrate proper use of the devices (drug pump and wearable device) will not be allowed to participate.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Infusion Site Reactions | 28 Days
  Local tolerability (infusion site evaluation) was assessed using the Infusion Site Assessment 2-part rating scale.
Number of Participants with Adverse Events | From first dose of study drug to 30 days after last dose of study drug (up to 2 months)
  Treatment emergent adverse events defined as any adverse event from the time of study drug administration until 30 days after discontinuation of study drug.
Percentage of Participants with Markedly Abnormal Vital Signs Values | 28 days
  Vital signs will be collected both supine and standing.
Columbia-Suicide Severity Rating Scale (C-SSRS) | 28 days
  The C-SSRS is an instrument designed to assess suicidal behavior and ideation.
Percentage of Participants with Potentially Clinically Significant Laboratory Values | 28 days
  Blood samples for serum chemistry tests will be collected following a minimum 8-hour fast.
Percentage of Participants with Potentially Clinically Significant Electrocardiogram (ECG) Results | 28 days
  A 12-lead ECG will be performed after the participant has been supine for at least 5 minutes.

SECONDARY OUTCOMES:
Plasma Concentrations of Levodopa | Days 1, 7, 14, 21, and 28
  Blood samples for pharmacokinetic assessment will be collected twice at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (12):
- United States (12):
  - Banner Sun Health Res Inst /ID# 165840, Sun City, Arizona
  - Loma Linda University /ID# 165592, Loma Linda, California
  - Univ CA, Irvine Med Ctr /ID# 165594, Orange, California
  - Compass Research /ID# 167329, Orlando, Florida
  - Univ Kansas Med Ctr /ID# 166280, Kansas City, Kansas
  - University of Kentucky Chandler Medical Center /ID# 164407, Lexington, Kentucky
  - University of Louisville /ID# 164997, Louisville, Kentucky
  - Washington University-School of Medicine /ID# 164412, St Louis, Missouri
  - NYU Langone Medical Center /ID# 164924, New York, New York
  - University of Cincinnati /ID# 165142, Cincinnati, Ohio
  - Cleveland Clinic Foundation /ID# 164413, Cleveland, Ohio
  - Neurology Consultants of Dallas /ID# 167116, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=M15-739#additional-resources-section